CLINICAL TRIAL: NCT07200310
Title: Hearing and Eustachian/Vestibular Functions in Hot Air Balloon Pilots: A Cross-sectional Matched-Control Study
Brief Title: Hearing/ET/Vestibular in Balloon Pilots
Acronym: FLIGHT-EAR
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Cappadoc-baloon-odio
Record Dates: First submitted 2025-09-13; First posted 2025-10-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss, Noise-Induced; Eustachian Tube Dysfunction; Vestibular Disorders; Occupational Exposure
Keywords: Hot-Air Balloon Pilots; Noise Exposure; Hearing Loss; Eustachian Tube Function; Vestibular Function; cVEMP; Otoacoustic Emissions (OAE); Acoustic Reflex; Occupational Health; Altitude / Barometric Pressure
MeSH Terms: conditions — Hearing Loss, Noise-Induced; Hearing Loss | interventions — Hearing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hot-Air Balloon Pilots: Licensed, professional and actively flying hot-air balloon pilots (≥18 years) with regular flight over the past 12 months (on average 5 days per week and at least 20 flights in month), not using any hearing-protection equipment, and typically each flying et least 60-90 minutes.
  Participants undergo a single non-invasive laboratory session including, tympanometry, tympanometry with maneuvers (Valsalva/Toynbee) for Eustachian tube function, pure-tone audiometry, otoacoustic emission (OAE) testing, acoustic reflex thresholds, and cervical vestibular evoked myogenic potential (cVEMP). No drugs, devices, or biospecimens are used.
  Interventions: Other: Non-invasive audiologic and vestibular assessments
- Control Group: Age (≥18 years) without occupational or recreational exposure to noise, altitude, or barometric pressure changes. Participants undergo the same single non-invasive laboratory session as the pilot group (tympanometry, pure-tone audiometry, OAE tests, acoustic reflex thresholds, and cVEMP). No drugs, devices, or biospecimens are used.
  Interventions: Other: Non-invasive audiologic and vestibular assessments

INTERVENTIONS:
Other: Non-invasive audiologic and vestibular assessments — standardized, single-session test battery performed in a sound-treated clinical laboratory. Procedures include tympanometry, tympanometry with simple maneuvers (Valsalva/Toynbee) for Eustachian tube function, pure-tone audiometry, otoacoustic emission (OAE) testing, acoustic reflex thresholds, and cervical vestibular evoked myogenic potentials (cVEMP) with EMG monitoring for adequate sternocleidomastoid activation. Testing is non-invasive, takes ~60 minutes, and is conducted under routine clinical practice conditions. No investigational drugs, devices, or biospecimens are used.
  Other Names: Audiologic and vestibular test battery; Hearing and balance function tests; Audiologic evaluations; Vestibular assessments

SUMMARY:
This study looks at whether working as a hot-air balloon pilot-being exposed to burner noise, changes in air pressure/temperature, and vertical acceleration-is linked to changes in hearing, Eustachian tube function, and vestibular (balance) function. Adult pilots from Cappadocia will be compared with adults who do not have these exposures.

Approximately 90 participants are expected to be enrolled For contextual exposure information, representative in-field noise measurements during balloon operations and basic flight parameters may be documented

Each participant will attend one visit (~60 minutes) in an ENT/audiology laboratory. After a short questionnaire and an ear exam (otoscopy), the following non-invasive tests will be performed: tympanometry; tympanometry with simple maneuvers (Valsalva/Toynbee) to evaluate Eustachian tube function (ΔTPP); pure-tone audiometry (including extended high frequencies); otoacoustic emission tests (TEOAE and DPOAE); acoustic (stapedius) reflex thresholds; and a brief cervical vestibular evoked myogenic potential (cVEMP) test. Symptom-triggered questionnaires will also be used: for participants reporting tinnitus, the Tinnitus Handicap Inventory (THI); for those reporting dizziness, the Berg Balance Scale (BBS).

No medications or blood tests are involved. Testing is safe and routinely used in clinical care. Risks are minimal (for example, temporary ear-canal pressure or brief dizziness). Testing will be stopped if any discomfort occurs. Personal information will be kept confidential, and results will be reported only in group form. Findings from this study may help improve occupational health guidance for hot-air balloon pilots.

DETAILED DESCRIPTION:
This study looks at whether working as a hot-air balloon pilot-being exposed to burner noise, changes in air pressure/temperature, and vertical acceleration-is linked to changes in hearing, Eustachian tube function, and vestibular (balance) function. Adult pilots from Cappadocia will be compared with adults who do not have these exposures.

Approximately 90 participants are expected to be enrolled For contextual exposure information, representative in-field noise measurements during balloon operations and basic flight parameters may be documented

Each participant will attend one visit (~60 minutes) in an ENT/audiology laboratory. This is a cross-sectional study with a single assessment visit. The following non-invasive tests will be performed

Tympanometry.

Acoustic (stapedius) reflex thresholds.

Tympanometry with simple maneuvers (Valsalva/Toynbee) to evaluate Eustachian tube function (pressure change in the middle ear) (ΔTPP).

Pure-tone audiometry (standard clinical frequencies and extended high frequencies).

Otoacoustic emission tests (OAE), including transient-evoked (TEOAE) and distortion-product (DPOAE), with analysis including high frequencies.

Cervical vestibular evoked myogenic potential (cVEMP) (a test of inner-ear balance reflexes), administered for all participants using a standardized protocol and EMG monitoring for adequate sternocleidomastoid activation.

Symptom-triggered questionnaires:

For participants reporting tinnitus, the Tinnitus Handicap Inventory (THI) will be administered.

For participants reporting dizziness, the Berg Balance Scale (BBS) will be administered.

Testing is non-invasive and performed in a sound-treated environment per routine clinical practice. If any discomfort (e.g., significant dizziness, pain, or elevated blood pressure) occurs, the relevant test is stopped and the participant may be withdrawn from testing at the investigator's discretion. For contextual exposure information, representative in-field noise measurements, air-pressure and altitude during balloon operations and basic flight parameters may be documented where available; these are not required for participation.

Data are recorded under coded study IDs and stored on secure institutional servers with access restricted to authorized study staff. Results will be reported in aggregate to protect confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (preferably 18-70).

Pilot group: Licensed, professional and actively flying hot-air balloon pilots with regular flight over the past 12 months (on average 5 days per week and at least 20 flights in month), not using any hearing-protection equipment, and typically each flying et least 60-90 minutes.

Control group: Adults without occupational or recreational exposure to significant pressure/altitude/noise (e.g., no mountaineering, scuba diving, or cabin crew duties).

Otoscopic suitability for testing (no tympanic membrane perforation; no active ear infection).

Exclusion Criteria:

* Acute upper respiratory tract infection (URTI) or otitis at the time of testing.,
* High noise exposure within the past 24-48 hours (e.g., concert, workshop).
* Tympanic membrane perforation; impacted cerumen that cannot be cleared; chronic suppurative otitis; presence of an active ventilation (tympanostomy) tube.
* History of otologic surgery.
* Menière's disease; significant otosclerosis; vestibular neuritis within the past 6 months; recent sudden hearing loss.
* Significant neurological disease or history affecting balance (e.g., multiple sclerosis, stroke).
* Use of ototoxic medications within the past 3 months (e.g., aminoglycosides, cisplatin).
* Contraindications to cVEMP testing (e.g., significant cervical pathology or prior cervical surgery, uncontrolled hypertension, suspected advanced carotid artery disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) in two cohorts: (1)(Hot-Air Balloon Pilots) licensed hot-air balloon pilots operating in the Cappadocia/Nevşehir region with ≥10 flights in the prior 12 months; and (2)(Controls) age-matched adults with no occupational or recreational exposure to significant noise, altitude, or barometric pressure variation (e.g., non-pilots, non-divers, non-cabin crew). Participants are healthy volunteers with otoscopic suitability (no perforation or active infection). Recruitment is via local pilot companies/registries and the surrounding community; all assessments occur at the SBÜ Gaziosmanpaşa Training and Research Hospital ENT/audiology laboratory (single-center). Planned enrollment: 45 pilots and 45 controls.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2025-09-04 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Eustachian Tube Function (ΔTPP after Valsalva/Toynbee) | At baseline, single visit (~5 minutes)
  Tympanometric middle-ear pressure change (ΔTPP in daPa) after maneuvers will be recorded. Impaired function defined as ΔTPP ≤15 daPa.
Distortion Product Otoacoustic Emission (DPOAE) amplitudes at 1-12 kHz | At baseline, single visit (~5 minutes)
  Mean DPOAE amplitudes at 1-12 kHz will be compared between hot-air balloon pilots and controls. Lower amplitudes are hypothesized in pilots with greater flight exposure.
Transient-Evoked Otoacoustic Emission (TEOAE) | At baseline, single visit (~5 minutes)
  Description: Mean TEOAE SNRs (dB) in half-octave bands from 1-4 kHz (and overall response/reproducibility %) will be compared between hot-air balloon pilots and controls. Lower SNRs are hypothesized in pilots with greater flight exposure.

SECONDARY OUTCOMES:
Tympanometry middle-ear pressure (TPP) and compliance | At baseline, single visit (~3 minutes)
  Description: Tympanometric peak pressure (TPP, daPa) and middle-ear compliance (ml) values will be obtained and compared between hot-air balloon pilots and controls. Abnormal or more negative TPP values are hypothesized in pilots with greater flight exposure, indicating possible Eustachian tube dysfunction.
Pure-Tone Audiometry thresholds | At baseline, single visit
  Air-conduction thresholds at standard clinical frequencies and high frequencies. Hypothesis: higher thresholds in pilots.
Cervical Vestibular Evoked Myogenic Potential (cVEMP) parameters | At baseline, single visit
  cVEMP amplitude and latency measured bilaterally. Hypothesis: altered responses in pilots.
Acoustic Reflex Thresholds | At baseline, single visit
  Lowest sound level (dB HL) eliciting stapedius reflex, when measurable.
In-field noise metrics during balloon operation (exploratory) | During balloon flight, single observation (~60-90 minutes)
  LAeq, LAFmax, and LCpeak recorded for contextual analysis. During flight observations (subset only)
Tinnitus Handicap Inventory (THI) score | Baseline, single visit
  Self-reported tinnitus-related handicap, total score (0-100).
Berg Balance Scale (BBS) score | Baseline, single visit
  Self-reported balance function, 14-item scale (0-56).

CONTACTS AND LOCATIONS:
Overall Officials: Ethem İlhan, MD, Principal Investigator — University of Health Sciences, Gaziosmanpaşa Training and Research Hospital (Istanbul, Turkey)
Locations (2):
- Turkey (Türkiye) (2):
  - Cappadocia Field Site (Göreme) - On-site assessments at hot-air balloon pilot companies, Nevşehir, Göreme
  - University of Health Sciences, Gaziosmanpaşa Training and Research Hospital, Department of Otorhinolaryngology-Head & Neck Surgery (ENT/Audiology Laboratory), Istanbul

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD). The informed consent and protocol do not authorize IPD sharing, and the cohort is small and identifiable (hot-air balloon pilots in a defined region), increasing re-identification risk. Per protocol, only aggregate, de-identified results will be reported; source data remain on secure institutional servers accessible only to the study team.

REFERENCES:
- [Result] Avci D, Sahin MI. Are the hearing and eustachian tube functions of the hot air balloon pilots disturbed? Auris Nasus Larynx. 2022 Aug;49(4):577-583. doi: 10.1016/j.anl.2021.11.002. Epub 2021 Nov 25. PMID 34840034
- [Result] Sahin Ceylan D, Sacli Y, Gultekin G, Avsar B, Ozver AG. Do Flights Affect Hearing in Hot Air Balloon Pilots? Am J Audiol. 2023 Nov 22:1-10. doi: 10.1044/2023_AJA-23-00126. Online ahead of print. PMID 37992408